CLINICAL TRIAL: NCT05067972
Title: A PHASE 1 DOSE ESCALATION AND EXPANSION STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETIC, PHARMACODYNAMIC, AND ANTITUMOR ACTIVITY OF PF-07260437 IN ADVANCED OR METASTATIC SOLID TUMORS
Brief Title: A Study of PF-07260437 in Advanced or Metastatic Solid Tumors
Acronym: C4431001
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Pfizer has made an internal business decision to not continue further development of PF-07260437. This decision was not due to major safety concerns or requests from any regulatory authorities.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4431001
Record Dates: First submitted 2021-09-24; First posted 2021-10-05 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Neoplasms; Endometrial Neoplasms; Breast Neoplasms
Keywords: Cancer of Endometrium; Cancer of the Endometrium; Carcinoma of Endometrium; Endometrial Cancer; Endometrial Carcinoma; Endometrium Cancer; Neoplasms, Endometrial; Cancer of Ovary; Cancer of the Ovary; Neoplasms, Ovarian; Ovarian Cancer; Ovary Cancer; Ovary Neoplasms; Breast Cancer; Breast Carcinoma; Breast Tumors; Cancer of Breast; Cancer of the Breast; Human Mammary Carcinoma; Malignant Neoplasm of Breast; Malignant Tumor of Breast
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Monotherapy dose escalation (Part 1) (Experimental): Participants will receive PF-07260437
  Interventions: Drug: PF-07260437
- Dose Expansion (Part 2A) - Tumor specific Arm A (Experimental): Participants will receive PF-07260437
  Interventions: Drug: PF-07260437; Diagnostic Test: B7-H4 IHC
- Dose Expansion (Part 2B) - Tumor specific Arm B (Experimental): Participants will receive PF-07260437
  Interventions: Drug: PF-07260437; Diagnostic Test: B7-H4 IHC
- Dose Expansion (Part 2C) - Tumor specific Arm C (Experimental): Participants will receive PF07260437
  Interventions: Drug: PF-07260437; Diagnostic Test: B7-H4 IHC

INTERVENTIONS:
Drug: PF-07260437 — B7-H4 x CD3 bi-specific mAb
  Other Names: B7-H4
Diagnostic Test: B7-H4 IHC — B7-H4 expression
  Arms: Dose Expansion (Part 2A) - Tumor specific Arm A; Dose Expansion (Part 2B) - Tumor specific Arm B; Dose Expansion (Part 2C) - Tumor specific Arm C

SUMMARY:
A study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and antitumor activity of PF-07260437, a B7-H4 x CD3 bispecific mAb, in participants aged ≥18 years of age with advanced or metastatic breast cancer, ovarian cancer or endometrial cancer. Adult participants with other advanced or metastatic high B7-H4 expressing tumors may be considered after discussion with and approval from sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Histological/cytological diagnosis of selected locally advanced or metastatic breast cancer, endometrial cancer and ovarian cancer
* Part 2A:In second line or more, participants with histological/cytological diagnosis of locally advanced or metastatic HR+ HER2- breast cancer showing high B7-H4 expression
* Part 2B: In second line or more participants with histological or cytological diagnosis of locally advance or metastatic HR+ Her2- breast cancer or triple negative breast cancer (TNBC) with no biomarker pre-selection
* Part 2C: In second line or more participants with histological diagnosis of locally advance or metastatic triple negative breast cancer with high B7-H4 expression
* Thyroid function within normal laboratory range; in participants with abnormal thyroid function if Free T4 is normal and participant is clinically euthyroid, participants is eligible

Exclusion Criteria:

* Participants with any active malignancy within 3 years prior to enrollment
* Participants with advanced/metastatic, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term (including participants with massive uncontrolled effusions [pleural, pericardial, peritoneal], pulmonary lymphangitis, and over 50% liver involvement).
* History of Grade ≥3 immune mediated adverse events (including liver function tests that where considered drug related and cytokine release syndrome) that was considered related to prior immune modulatory therapy (eg, immune checkpoint inhibitors, co stimulatory agents, etc.) and required immunosuppressive therapy within 1 year of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- United States (12):
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - Moffitt Cancer Center at McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - The University of Chicago Medicine Center of Advanced Care Orland Park, Orland Park, Illinois
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - NEXT Oncology, San Antonio, Texas
  - Swedish Cancer Institute Edmonds Campus, Edmonds, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Mountlake, Seattle, Washington
- Puerto Rico (3):
  - Pan American Center for Oncology Trials, LLC, Rio Piedras
  - Pan American Center for Oncology Trials- Hospital Oncologico, Rio Piedras
  - Pan American Center for Oncology Trials, Rio Piedras

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4431001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The decision to terminate the study was made on 27 July 2023, due to strategic reasons. By the time of study termination, Part 2 of the study has not been initiated. Therefore, only results from Part 1 are presented.
Groups:
- PF-07260437 100 ug SC Q2W: Participants with locally advanced or metastatic breast cancer (BrCa), ovarian cancer (OvCa) or endometrial cancer received PF-07260437 100 microgram (ug) by subcutaneous (SC) injection every 2 weeks (Q2W) in 28-day cycles (on Days 1 and 15) until the participant met one of the study intervention discontinuation criteria.
- PF-07260437 300 ug SC Q2W: Participants with locally advanced or metastatic BrCa, OvCa or endometrial cancer received PF-07260437 300 ug by SC injection Q2W in 28-day cycles (on Days 1 and 15) until the participant met one of the study intervention discontinuation criteria.
- PF-07260437 500 ug SC Q2W: Participants with locally advanced or metastatic BrCa, OvCa or endometrial cancer received PF-07260437 500 ug by SC injection Q2W in 28-day cycles (on Days 1 and 15) until the participant met one of the study intervention discontinuation criteria.
- PF-07260437 200 ug (Priming) + 500 ug SC Q2W: Participants with locally advanced or metastatic BrCa, OvCa or endometrial cancer received PF-07260437 priming dose of 200 ug on C1D1 (Cycle 1 Day 1) and full/maintenance dose of 500 ug on C1D15 and afterwards by SC injection Q2W in 28-day cycles (Days 1 and 15) until the participant met one of the study intervention discontinuation criteria.
- PF-07260437 200 ug (Priming) + 800 ug SC Q2W: Participants with locally advanced or metastatic BrCa, OvCa or endometrial cancer received PF-07260437 priming dose of 200 ug on C1D1 and full/maintenance dose of 800 ug on C1D15 and afterwards by SC injection Q2W in 28-day cycles (Days 1 and 15) until the participant met one of the study intervention discontinuation criteria.
- PF-07260437 100 ug (First Priming) + 300 ug (Second Priming) + 800 ug SC Q2W: Participants with locally advanced or metastatic BrCa, OvCa or endometrial cancer received PF-07260437 first priming dose of 100 ug on C1D1, second priming dose of 300 ug on C1D8, and full/maintenance dose of 800 ug on C1D15 and afterwards by SC injection Q2W in 28-day cycles (Days 1 and 15) until the participant met one of the study intervention discontinuation criteria.
- PF-07260437 200 ug (Priming) + 1600 ug SC Q2W: Participants with locally advanced or metastatic BrCa, OvCa or endometrial cancer received PF-07260437 priming dose of 200 ug on C1D1 and full/maintenance dose of 1600 ug on C1D15 and afterwards by SC injection Q2W in 28-day cycles (Days 1 and 15) until the participant met one of the study intervention discontinuation criteria.
Period: Part 1: Treatment
Arm/Group | PF-07260437 100 ug SC Q2W | PF-07260437 300 ug SC Q2W | PF-07260437 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 800 ug SC Q2W | PF-07260437 100 ug (First Priming) + 300 ug (Second Priming) + 800 ug SC Q2W | PF-07260437 200 ug (Priming) + 1600 ug SC Q2W
Started | 3 | 4 | 4 | 6 | 4 | 4 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 4 | 6 | 4 | 4 | 5
Not completed — Global Deterioration of Health Status | 0 | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Progressive Disease | 3 | 3 | 4 | 2 | 3 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 1
Period: Part 1: Follow-up
Arm/Group | PF-07260437 100 ug SC Q2W | PF-07260437 300 ug SC Q2W | PF-07260437 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 800 ug SC Q2W | PF-07260437 100 ug (First Priming) + 300 ug (Second Priming) + 800 ug SC Q2W | PF-07260437 200 ug (Priming) + 1600 ug SC Q2W
Started | 1 | 3 | 4 | 4 | 2 | 3 | 4
Completed | 0 | 1 | 3 | 3 | 1 | 1 | 2
Not Completed | 1 | 2 | 1 | 1 | 1 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 1 | 2 | 1 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-07260437 100 ug SC Q2W | PF-07260437 300 ug SC Q2W | PF-07260437 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 800 ug SC Q2W | PF-07260437 100 ug (First Priming) + 300 ug (Second Priming) + 800 ug SC Q2W | PF-07260437 200 ug (Priming) + 1600 ug SC Q2W | Total
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 4 | 4 | 5 | 30
Age, Continuous [Median (Full Range); unit: Years] | 58 [44 to 65] | 66 [60 to 73] | 58 [52 to 66] | 58 [41 to 75] | 67 [56 to 73] | 63.5 [58 to 69] | 60 [47 to 67] | 61 [41 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 6 | 4 | 4 | 5 | 30
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 3 | 1 | 2 | 1 | 9
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 3 | 2 | 4 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 3 | 4 | 4 | 5 | 2 | 3 | 4 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs) in Dose Escalation - Part 1
Description: Any of the following treatment-related adverse events (AEs) occurring during the DLT observation period were classified as DLTs: Hematological DLTs: neutropenia Grade (G) 4, febrile neutropenia, ≥G3 for >7d (days), G3 with infection; thrombocytopenia G4, G3 with bleeding or requiring platelet transfusion; anemia G4, G3 requiring blood transfusion. Non-hematologic: hepatic toxicity; ≥G3 fatigue for ≥5d, ≥G3 nausea/vomiting or diarrhea for ≥3d, ≥G3 cytokine release syndrome (CRS) of any duration/QTcF prolongation/anaphylaxis, G5 AE without clear reason; immune-related (ir)AE: ≥G4 irAEs/colitis, G3/4 non-infectious pneumonitis, G2 pneumonitis not resolved to ≤G1 within 3d of the initiation of max supportive care. Severity of AEs were graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, with the exception of CRS, which were graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) CRS Consensus Grading for CRS.
Time Frame: The first dose of the study intervention (C1D1) through Day 28 for participants without a priming dose or through Day 42 for participants with a priming dose.
Population: DLT evaluable set included all enrolled participants who had at least 1 dose of study intervention and either experienced DLT or did not have major protocol deviations during the DLT observation period.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07260437 100 ug SC Q2W | PF-07260437 300 ug SC Q2W | PF-07260437 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 800 ug SC Q2W | PF-07260437 100 ug (First Priming) + 300 ug (Second Priming) + 800 ug SC Q2W | PF-07260437 200 ug (Priming) + 1600 ug SC Q2W
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 2 | 2
Participants | 0 | 0 | 1 | 0 | 0 | 2 | 1

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) - Part 1
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAE was defined as any AE that occurred from first dose of study intervention to either last dose of study treatment + 90 days, start of new anti-cancer therapy, or completion in study as determined by disposition, whichever was earliest. A serious AE (SAE) was defined as any untoward medical occurrence that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, persistent disability/incapacity, or was a congenital anomaly/birth defect. AEs were graded by the investigator according to CTCAE v5.0.
Time Frame: Baseline (Day 1 of dosing ) through 4 week follow-up, up to 35.1 weeks
Population: All enrolled participants who received at least one dose of study intervention were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07260437 100 ug SC Q2W | PF-07260437 300 ug SC Q2W | PF-07260437 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 800 ug SC Q2W | PF-07260437 100 ug (First Priming) + 300 ug (Second Priming) + 800 ug SC Q2W | PF-07260437 200 ug (Priming) + 1600 ug SC Q2W
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 4 | 4 | 5
Participants
  Participants with all-causality TEAEs | 3 | 4 | 4 | 6 | 4 | 4 | 5
  Participants with treatment-related TEAEs | 3 | 4 | 4 | 5 | 4 | 4 | 5
  Participants with all-causality treatment-emergent SAEs | 0 | 2 | 1 | 5 | 1 | 3 | 2
  Participants with treatment-related treatment-emergent SAEs | 0 | 1 | 1 | 3 | 1 | 3 | 2
  Participants with maximum Grade 3 or 4 TEAEs - all-causality | 1 | 3 | 3 | 4 | 0 | 4 | 5
  Participants with maximum Grade 3 or 4 TEAEs - treatment related | 1 | 3 | 3 | 5 | 0 | 4 | 5
  Participants with maximum Grade 5 TEAEs - all-causality | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Participants with maximum Grade 5 TEAEs - treatment related | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with immune-related TEAEs - all-causality | 1 | 0 | 0 | 0 | 1 | 1 | 1
  Participants with immune-related TEAEs - treatment-related | 1 | 0 | 0 | 0 | 1 | 1 | 1

3. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities - Part 1
Description: Laboratory parameters included: hematology (hemoglobin, hematocrit, red blood cell, platelet and white blood cell count, neutrophils, eosinophils, monocytes, basophils and lymphocytes), chemistry (blood urea nitrogen, creatinine, sodium, potassium, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein and serum pregnancy test [for all female participants]) and urine (urine pregnancy test [for all female participants]). Clinical significance of laboratory parameters was determined at the investigator's discretion.
Time Frame: Baseline through up to 35.1 weeks
Population: All enrolled participants who received at least one dose of study intervention were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07260437 100 ug SC Q2W | PF-07260437 300 ug SC Q2W | PF-07260437 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 800 ug SC Q2W | PF-07260437 100 ug (First Priming) + 300 ug (Second Priming) + 800 ug SC Q2W | PF-07260437 200 ug (Priming) + 1600 ug SC Q2W
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Immune-Related Adverse Events (irAEs)
Description: irAEs included gastrointestinal (ie, diarrhea/colitis), dermatological (ie, rash), pulmonary (ie, pneumonitis), hepatic (ie, liver test elevation), renal (ie, creatinine increased), cardiac (ie, myocarditis), endocrine (ie, endocrine disorder), and other toxicities.
Time Frame: Day 1 up to 90 days after the last dose of study intervention (Day 246 [C9D15]), up to approximately 336 days
Population: All enrolled participants who receive at least 1 dose of study intervention were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07260437 100 ug SC Q2W | PF-07260437 300 ug SC Q2W | PF-07260437 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 800 ug SC Q2W | PF-07260437 100 ug (First Priming) + 300 ug (Second Priming) + 800 ug SC Q2W | PF-07260437 200 ug (Priming) + 1600 ug SC Q2W
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 4 | 4 | 5
Participants | 1 | 0 | 0 | 0 | 1 | 1 | 1

5. Secondary Outcome: Number of Participants by Categories of Anti-Drug Antibody (ADA) Against PF-07260437
Description: Number of participants with positive ADA against PF-07257876 were summarized for each treatment arm. A participant had treatment-induced ADA response if he/she had negative or missing ADA at baseline and ≥1 post-treatment ADA positive titer. A participant had treatment-boosted ADA response if he/she had positive titer at baseline and a ratio of ≥4 in titer (dilution) to baseline in ≥1 post-treatment sample.
Time Frame: On Day 1 of Cycle 1, 2, 3. From Cycle 4 onwards: collection on Day 1 of every 3 cycles (C4D1, C7D1, etc.) until end-of-treatment visit, up to 35.1 weeks.
Population: The immunogenicity analysis set included all enrolled participants who received at least 1 dose of study treatment and had at least 1 sample tested for ADA.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07260437 100 ug SC Q2W | PF-07260437 300 ug SC Q2W | PF-07260437 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 800 ug SC Q2W | PF-07260437 100 ug (First Priming) + 300 ug (Second Priming) + 800 ug SC Q2W | PF-07260437 200 ug (Priming) + 1600 ug SC Q2W
Number analyzed (Participants) | 3 | 4 | 4 | 5 | 3 | 3 | 4
Participants
  Participant with treatment-induced ADA response | 1 | 2 | 0 | 1 | 0 | 1 | 2
  Participant with treatment-boosted ADA response | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Single Dose: Maximal Concentration (Cmax)
Description: Maximum observed serum concentration following single dose of PF-07260437. The multiple dose PK samples were not collected due to dose interruption or discontinuation. The PK sampling schedule was designed to evaluate the dosing interval of 2 weeks. Since the 100/300/800 group received the second dose (300 ug) only 1 week after the first dose. The PK parameters were not calculable.
Time Frame: Day 1 pre-dose, 1, 4, 8, 24, 48 and 168 hours post-dose, till Day 15 pre-dose in Cycle 1
Population: All enrolled participants treated who did not have protocol deviations influencing PK assessment and had sufficient information to estimate at least 1 of the PK parameters of interest. Participants with ≤3 sampling points or missing PK samples on day 14 were excluded. Participants in 200/500, 200/800, 200/1600 groups received the same dose on Day 1, and therefore, were combined for single dose (200 ug) PK to increase the sample size and provide more confidence to the estimate.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- PF-07260437 200 ug: The group of 200 ug dose includes participants who received an identical priming dose (200 ug) from 200/500, 200/800, and 200/1600 Q2W dose groups.
Arm/Group | PF-07260437 100 ug SC Q2W | PF-07260437 200 ug | PF-07260437 300 ug SC Q2W | PF-07260437 500 ug SC Q2W | PF-07260437 100 ug (First Priming) + 300 ug (Second Priming) + 800 ug SC Q2W
Number analyzed (Participants) | 3 | 11 | 3 | 3 | 0
ng/mL | 5.75 (31.9) | 16.2 (69.9) | 37.2 (22.5) | 33.0 (45.2) |

7. Secondary Outcome: Single Dose: Area Under the Curve (AUCtau)
Description: Area under the plasma concentration-time profile from time 0 to time tau (τ), the dosing interval following single dose of PF-07260437. The multiple dose PK samples were not collected due to dose interruption or discontinuation. The PK sampling schedule was designed to evaluate the dosing interval of 2 weeks. Since the 100/300/800 group received the second dose (300 ug) only 1 week after the first dose. The PK parameters were not calculable.
Time Frame: Day 1 pre-dose, 1, 4, 8, 24, 48 and 168 hours post-dose, till Day 15 pre-dose in Cycle 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*day/mL
Arm/Group | PF-07260437 100 ug SC Q2W | PF-07260437 200 ug | PF-07260437 300 ug SC Q2W | PF-07260437 500 ug SC Q2W | PF-07260437 100 ug (First Priming) + 300 ug (Second Priming) + 800 ug SC Q2W
Number analyzed (Participants) | 3 | 11 | 3 | 3 | 0
ng*day/mL | 62.1 (21.2) | 148 (74.0) | 424 (25.1) | 332 (37.8) |

8. Secondary Outcome: Single Dose: Time to Maximal Plasma Concentration (Tmax)
Description: Time to maximal plasma concentration following single dose of PF-07260437. The multiple dose PK samples were not collected due to dose interruption or discontinuation. The PK sampling schedule was designed to evaluate the dosing interval of 2 weeks. Since the 100/300/800 group received the second dose (300 ug) only 1 week after the first dose. The PK parameters were not calculable.
Time Frame: Day 1 pre-dose, 1, 4, 8, 24, 48 and 168 hours post-dose, till Day 15 pre-dose in Cycle 1
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | PF-07260437 100 ug SC Q2W | PF-07260437 200 ug | PF-07260437 300 ug SC Q2W | PF-07260437 500 ug SC Q2W | PF-07260437 100 ug (First Priming) + 300 ug (Second Priming) + 800 ug SC Q2W
Number analyzed (Participants) | 3 | 11 | 3 | 3 | 0
days | 7.00 [7.00 to 7.00] | 7.00 [7.00 to 7.00] | 7.00 [7.00 to 7.00] | 7.00 [7.00 to 7.00] |

ADVERSE EVENTS:
Time Frame: Baseline through up to 35.1 weeks
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, persistent disability/incapacity, or was a congenital anomaly/birth defect.
Arm/Group | PF-07260437 100 ug SC Q2W | PF-07260437 300 ug SC Q2W | PF-07260437 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 500 ug SC Q2W | PF-07260437 200 ug (Priming) + 800 ug SC Q2W | PF-07260437 100 ug (First Priming) + 300 ug (Second Priming) + 800 ug SC Q2W | PF-07260437 200 ug (Priming) + 1600 ug SC Q2W
All-Cause Mortality (participants affected / at risk) | 1/3 | 3/4 | 1/4 | 2/6 | 1/4 | 0/4 | 1/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/4 | 1/4 | 5/6 | 1/4 | 3/4 | 2/5
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 4/4 | 6/6 | 4/4 | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-07260437 100 ug SC Q2W (N=3) | PF-07260437 300 ug SC Q2W (N=4) | PF-07260437 500 ug SC Q2W (N=4) | PF-07260437 200 ug (Priming) + 500 ug SC Q2W (N=6) | PF-07260437 200 ug (Priming) + 800 ug SC Q2W (N=4) | PF-07260437 100 ug (First Priming) + 300 ug (Second Priming) + 800 ug SC Q2W (N=4) | PF-07260437 200 ug (Priming) + 1600 ug SC Q2W (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07260437 100 ug SC Q2W (N=3) | PF-07260437 300 ug SC Q2W (N=4) | PF-07260437 500 ug SC Q2W (N=4) | PF-07260437 200 ug (Priming) + 500 ug SC Q2W (N=6) | PF-07260437 200 ug (Priming) + 800 ug SC Q2W (N=4) | PF-07260437 100 ug (First Priming) + 300 ug (Second Priming) + 800 ug SC Q2W (N=4) | PF-07260437 200 ug (Priming) + 1600 ug SC Q2W (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 3 | 1 | 2 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 1 | 1 | 1
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 1 | 3 | 3 | 3 | 2
Influenza like illness (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 2 | 2 | 1 | 2 | 2 | 2 | 2
Localised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 2
Cytokine release syndrome (Immune system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 2
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 3 | 4 | 2 | 4 | 5
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anion gap increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 4 | 4 | 2 | 4 | 4
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 3 | 4 | 1 | 4 | 4
Blood bilirubin increased (Investigations) | 0 | 2 | 1 | 2 | 0 | 4 | 5
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Electrocardiogram ST-T segment abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 1
Lung diffusion test decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 2 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 3 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 2 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight fluctuation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 1 | 2 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 0 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The decision to terminate the study was made on 27 Jul 2023, due to strategic reasons. The multiple dose PK samples were not collected due to dose interruption or discontinuation. By the time of study termination, Part 2 of the study has not been initiated. Therefore, no data have been collected for Part 2 and corresponding endpoints were not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT05067972/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT05067972/SAP_001.pdf